CLINICAL TRIAL: NCT03296709
Title: Preformed Pediatric Crown Zirconia Versus Preformed Pediatric Metal Crown PPC Z-M
Brief Title: Preformed Pediatric Crown Zirconia Versus Preformed Pediatric Metal Crown
Acronym: PPC Z-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-PP-08
Record Dates: First submitted 2017-07-28; First posted 2017-09-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Tooth Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Split mouth design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPC m (Active Comparator)
  Interventions: Device: PPC m
- PPC z (Experimental)
  Interventions: Device: PPC z

INTERVENTIONS:
Device: PPC z — Installation of a preformed pediatric zircona crown
  Arms: PPC z
Device: PPC m — Installation of a preformed pediatric metal crown
  Arms: PPC m

SUMMARY:
Preformed metal pediatric crowns (PPCm) are currently considered the best method of restoring Primary molars affected by severe carious lesions compared to restorations made with various restorative materials (amalgams, composites, CVI-based materials). Due to their unsightly appearance, denounced by many parents, more aesthetic zirconia (PPCz) preformed pediatric crowns have been recently marketed. In the absence of an evaluation of the latter, this multi-center split-mouth two-year randomized clinical trial (RCT) proposes to to investigate the effectiveness of PPCz for the management of dental caries or structural anomalies. More specifically, the primary objective of this RCT is to assess in primary molars the success of PPCz in comparison with PPCm. The control treatment will be PPCm since this is the standard crown option.

One hundred children and one aged at least 4 years must be recruited in ninedepartments of Pediatric Dentistry in the university hospitals of Bordeaux, Lille, Nancy, Nantes, Nice, Paris 1&2, Strasbourg and Toulouse. They will be included if they have two similar primarymolars of the same arch (for example first right and left maxillary primary molars ) and equally affected, to be crowned. The two types of crowns to be used in the same child, PPCm(3M Espe) and PPCz(Ezpédo), will be affected by randomization using a computerized and centralized system: primary molars will first be allocated to PPCm and, one to two weeks later, the contralateral primary molar will be restored by PPCz. The children will be checked every 6 months for a period of 2 years after the placement of the two types of crowns . During these four control visits, primary and secondary outcomes will be assessed clinically and radiographically. The primary outcome is the success of the treatment defined by the absence of major failure. A composite measure of signs and symptoms leading to diagnosis of irreversible pulpitis or periradicular periodontitis will be used to define major failure (pain, pulp infection, dental abscess, periradicular pathology visible on radiograph). The secondary outcomes are parental and child satisfaction (size, form and color), retention and fracture of the PPC, the wear of the antagonist tooth, the gingival state near PPC using the indices Löe and Silness to record plaque index (PI), gingival index (GI) and depth of the pocket (DI) on the crowned tooth and the two adjacent ones. Each center has a trained and / or calibrated operator and evaluator.

ELIGIBILITY:
Inclusion Criteria:

* Children of at least 4 years of good general health (ASAI or II),
* Child with at least two temporary molars of the same type, 1st or 2nd molar, contralateral (fractional mouth), meeting the following criteria:

The two temporary molars are affected by a cavitary carious lesion or a hypoplastic defect of at least 2 faces,

* the two temporary molars of the pair (54-64, 55-65, 74-84 or 75-85), should or should not be subjected to pulpotomy prior to the realization of the CPP,
* the two molars must have an antagonistic tooth.

  * Consent of parents (legal guardians) and child,
  * Child and parents (legal guardians) speaking French,
  * Child covered by his parents' social security cover,
  * Child cooperating in the vigilant or sedated state (cooperation evaluated with a Venham score 0, 1, 2).

Exclusion Criteria:

* Child who does not cooperate in care under vigil or under conscious sedation, who must therefore be treated under general anesthesia.
* Child allergic to local anesthetics, chromium or nickel. Exclusion dental criteria
* Primary molar whose physiological exfoliation will appear within 24 months or pimary molar with a root resorption of more than a third of the radicular length.
* Severely decayed PM prohibiting the retention and the sealing of the restoration.
* Primary molar with exposed cement or with evidence of swelling in the surrounding tissues
* Molar with spontaneous pain.
* Primary molar in infraclusion.
* Primary molar whose radiographic examination reveals a widening of the desmodontal space, the presence of radiolucent image on the root furcation and/or apices, internal or external resorption

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
clinical and radiographique observations | 2 years
  Success of the treatment defined by the absence of major failure. A composite measure of signs and symptoms leading to diagnosis of irreversible pulpitis or periradicular periodontitis will be used to define major failure (pain, pulp infection, dental abscess, periradicular pathology visible on radiograph

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHRU Lille, Lille
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHU Stransbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Cazaux S, Aiem E, Velly AM, Muller-Bolla M. Preformed pediatric zirconia crown versus preformed pediatric metal crown: study protocol for a randomized clinical trial. Trials. 2019 Aug 24;20(1):530. doi: 10.1186/s13063-019-3559-1. PMID 31445509